CLINICAL TRIAL: NCT06743724
Title: Clinical Study of Repeated Transcranial Magnetic Stimulation(rTMS) for Maternal Care Impairment (MCI)
Brief Title: Repeated Transcranial Magnetic Stimulation Relieves Maternal Care Impairment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.2024-117
Record Dates: First submitted 2024-12-07; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Maternal Care Patterns; Repetitive Transcranial Magnetic Stimulation (rTMS); Functional Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-score group (Experimental): The low-score group received rTMS at 1 Hz for 20 minutes per session, once daily, for a duration of 2 weeks.
  Interventions: Device: repeated transcranial magnetic stimulation treatment

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation treatment — Patients with low score of Maternal Care Rating Scale received repetitive transcranial magnetic stimulation at 1 Hz/s for 20 minutes for 2 week.

SUMMARY:
Objective: To evaluate the overall efficacy of repetitive transcranial magnetic stimulation (rTMS) in the treatment of maternal care impairment and to explore the central mechanism of rTMS for maternal care impairment.

Methods: Fifty participants meeting the inclusion criteria were divided into high-score and low-score groups based on the Maternal Care Rating Scale (MCRS). Participants in the low-score group received rTMS treatment (1 Hz, 20 minutes per session, once daily) for two weeks. Functional magnetic resonance imaging (fMRI) and MCRS assessments were conducted both before and after the treatment to evaluate changes. Additionally, in the high-score group, fMRI was used to assess functional changes in specific brain regions.

DETAILED DESCRIPTION:
A substantial body of literature has reported that repetitive transcranial magnetic stimulation (rTMS) can alleviate negative emotions. The underlying mechanisms include its ability to modulate cortical excitability, enhance cerebral blood flow and metabolism, regulate neurotransmitter and gene expression, and promote neuroplastic changes in the nervous system.

Methods:

1. Fifty recruited volunteers were divided into high-score and low-score groups based on the Maternal Care Rating Scale (MCRS). Functional magnetic resonance imaging (fMRI) was used to assess differences in brain function between the two groups.
2. The low-score group underwent a two-week intervention with repetitive transcranial magnetic stimulation (rTMS) (1 Hz, 20 minutes per session, once daily). The MCRS served as the primary outcome measure to evaluate treatment efficacy. Additionally, fMRI was performed to compare pre- and post-treatment changes in brain function. The functional magnetic resonance data of both the high-score and low-score groups were analyzed using the amplitude of low-frequency fluctuation (ALFF) method and the regional homogeneity (ReHo) method to identify differences in brain function. For the low-score group, changes in ALFF and ReHo values in specific brain regions before and after treatment were compared. These changes were correlated with the improvement values of the clinical observation index to identify target brain areas that mediate the effects of rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers.
* Aged between 18 and 45 years.
* No pharmacological treatment (excluding emergency treatment) for at least 2 weeks prior to the start of treatment; cannot be enrolled in other clinical trials simultaneously.
* Voluntarily sign the informed consent form and willingly participate in the clinical study.

Exclusion Criteria:

* Age below 18 years or above 45 years.
* Unmarried, nulliparous women.
* Individuals with severe liver, kidney, hematological diseases, cardiovascular diseases, or other conditions that significantly affect cognitive function.
* Participants with a clear history of organic diseases, or systemic conditions such as diabetes, hyperthyroidism, etc.
* Participants undergoing other treatments or taking medications that may interfere with the outcome assessment.
* Pregnant women, breastfeeding women, or women within six months postpartum.
* Individuals with severe needle phobia, metal allergies, or allergic conditions, or those with a cardiac pacemaker.
* Participants who do not comply with random group assignment or have unstable tendencies such as poor adherence.
* Individuals currently participating in other research studies.
* Individuals unwilling to sign the informed consent form.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Maternal Care Rating Scale | 1 week of treatment
  The Maternal Care Rating Scale (MCRS) is a tool designed to assess and evaluate the quality of maternal care, including aspects of maternal behavior, emotional responses, and caregiving abilities. It focuses on the mother's ability to engage in positive, nurturing, and responsive interactions with her child. The scale can help identify variations in maternal care, such as maternal sensitivity, emotional support, and overall caregiving competence. In research, it is often used to measure the effectiveness of interventions aimed at improving maternal behavior or addressing maternal deficits, such as maternal care impairment (MCI).

CONTACTS AND LOCATIONS:
Overall Officials: Guangyin Xu, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China, China

IPD SHARING:
Plan to Share IPD: No
This clinical research protocol is just beginning to be studied at this time and sharing is not recommended at this time.